CLINICAL TRIAL: NCT00171288
Title: Efficacy and Safety Study of Fluvastatin and Ezetimibe Combined Versus Fluvastatin Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CXUO320BES03
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia, ezetimibe, inflammatory markers, fluvastatin
MeSH Terms: conditions — Dyslipidemias | interventions — Fluvastatin; Ezetimibe

INTERVENTIONS:
Drug: fluvastatin, ezetimibe

SUMMARY:
The objective of this study is to assess the effect of the combination treatment on C-reactive protein and inflammatory markers as well as the safety and tolerability in a Spanish population

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 Primary hypercholesterolemia Signed informed consent

Exclusion Criteria:

* Patients involved in clinical trials 3 months prior to inclusion Patients treated with drugs specified in protocol Fertile women not using contraceptive methods

Other protocol defined in and exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2003-08; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in low density lipoprotein cholesterol after 12 weeks

SECONDARY OUTCOMES:
Change from baseline in total triglyceride, high density lipoprotein cholesterol, and composition of low density lipoprotein cholesterol after 12 weeks
Change from baseline in circulating marker of inflammation after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Madrid, Spain